CLINICAL TRIAL: NCT00580164
Title: The Role of Splinting in Fingertip Injuries
Status: Withdrawn | Type: Observational
Why Stopped: Very few subjects were enrolled. Therefore, the study was terminated.
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, David C. Ring, MD, Principal Investigator, Massachusetts General Hospital
Other Study IDs: 2006-p000239
Record Dates: First submitted 2007-12-20; First posted 2007-12-24 (Estimated); Last update posted 2015-12-30 (Estimated); Status verified 2015-12

CONDITIONS: Injury Distal to Flexor and Extensor Tendon Insertions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Splint
- 2: No Splint

SUMMARY:
This study is attempting to understand whether or not splinting after a fingertip injury improves recovery.

ELIGIBILITY:
Inclusion Criteria:

* injury distal to flexor and extensor tendon insertions
* crush, avulsion, amputation, or penetrating injury to the fingertip
* isolated injury, within two weeks

Exclusion Criteria:

* operative fixation required
* unable to participate in rehab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Orthopaedic Hand Clinic
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2006-01; Primary Completion 2010-05 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
DASH questionnaire, Grip strength, and Range of Motion | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: David C Ring, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Mass General Hospital, Boston, Massachusetts, United States